CLINICAL TRIAL: NCT06083389
Title: The Role of Kabat Rehabilitation Technique Versus Conventional Physical Therapy Along With Electrical Stimulation in Treatment of Bell's Palsy
Brief Title: Kabat Rehabilitation Technique Versus Conventional Physical Therapy in Treatment of Bell's Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Aya Hassan AbdelAzeem Ahmed, assistant lecturer at faculty of medicine Minia university, Minia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rehabilitation of facial balsy
Record Dates: First submitted 2023-03-23; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Bell's Palsy
Keywords: rehabilitation facial palsy
MeSH Terms: conditions — Bell Palsy | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional technique of facial exercises along with electrical stimulation of facial muscles. (Active Comparator): facial muscle exercise active exercises will be initiated, which is performed in front of a mirror in sitting position. The patient will be instructed for activities like blowing air in the mouth, nasal flaring, smiling, raising and frowning of the eyebrows, opening and closing of the eye, clenching of the teeth and holding straw in mouth, suck and blow out air, show as if blowing a balloon for 20 minutes each session, for 3 sessions/ week for 6 weeks.
  Interventions: Device: electrotherapy
- Kabat technique arm along with stimulation of facial muscles. (Active Comparator): During the Kabat rehabilitation session, the patients will perform specific diagonal and spiral movements, involving the following three muscle fulcrums:
  * Upper fulcrum: includes the frontalis, corrugator & orbicularis oculi muscles.
  * Intermediate fulcrum: includes the common elevator muscle of the upper lip and nasalis.
  * Lower fulcrum: includes the risorius, zygomaticus major, the orbicularis oris and buccinator. (Khanzada et al., 2018).
  The manipulation of these three fulcra will be carried out by utilizing contralateral contraction and the basic proprioceptive stimulation comprising stretching, maximal resistance, manual contact and verbal input.
  Kabat sessions will be 3 sessions / week for 6 weeks.
  Interventions: Behavioral: kabat technique for rehabilitation of facial palsy; Device: electrotherapy

INTERVENTIONS:
Behavioral: kabat technique for rehabilitation of facial palsy — To evaluate the comparative effectiveness of the Kabat rehabilitation technique with conventional physical therapy along with electrical stimulation in both, for reducing facial disability in patients with Bell's palsy.
  Arms: Kabat technique arm along with stimulation of facial muscles.
Device: electrotherapy — electrical stimulation of facial nerve supplied muscles.3 sessions per week.

SUMMARY:
To evaluate the comparative effectiveness of the Kabat rehabilitation technique with conventional physical therapy along with electrical stimulation in both, for reducing facial disability in patients with Bell's palsy.

To assess the prognosis of patients with Bell's palsy, using the assay of serum level of ischemia-modified albumin, high-frequency ultrasonography (HFUS), and electrophysiological studies of the facial nerve.

DETAILED DESCRIPTION:
Bell's Palsy (BP), named after the Scottish anatomist and surgeon Sir Charles Bell who first described it, is a disease that occurs as a result of idiopathic usually unilateral, and isolated seventh cranial nerve (facial nerve) paralysis, leading to an inability to control the facial muscles on the affected side without a known cause . Bell's Palsy is the most common acute mononeuropathy, accounting for approximately 60%-75% of all cases of unilateral facial paralysis . The incidence of BP ranges from 11.5 to 40.2 in 100,000 cases. Although it may influence all ages, it is more commonly seen between 15 and 45 years old .

The imbalance between pro-oxidants and antioxidants, if not deactivated by the cellular antioxidant system, results in oxidative stress status. Reactive oxygen species (ROS) derived from ischaemic events can generate products leading to cellular deregulation. Excess of these species can react with cellular macromolecules and results in lipid peroxidation, nucleic acid damages and protein modifications .

Systemic markers of oxidative stress include ischemia-modified albumin (IMA). When tissue ischemia occurs, a newly formed albumin called IMA is produced. It is suggested that BP patients have higher serum levels of IMA due to excess ROS and so oxidative stress status providing information about the relationship between oxidative stress status and BP .

Electro neurophysiology is the main diagnostic and prognostic tool in peripheral neuropathy. Facial nerve electrodiagnostic is a well-established and important tool for decision-making in patients with facial nerve diseases. Electro neurophysiological analyses of the facial nerve and facial muscles can assist in diagnosis, assess the lesion severity, and it is a valuable tool for predicting recovery.

Ultrasonography has increasingly been used to investigate neuromuscular disorders. It enables real-time imaging acquisition, is easily accessible, and can be used at the bedside. Furthermore, it can be used to diagnose and predict prognosis in neuromuscular disorders, as well as to assess structural lesions in nerves. With advances in image resolution, some cranial nerves, including the facial nerve, have also become accessible to ultrasonographic imaging. Neuromuscular ultrasound may be helpful in the diagnosis and disease prognosis. Serial ultrasonographic scanning of the facial nerve from disease onset until recovery may also help advance this promising technique.

Bell's palsy is commonly treated by various physical therapy strategies. Physiotherapy treatment for Bell's palsy includes kinesiotherapy, massage therapy, cryotherapy and electrotherapy. Electrical stimulation (ES) of paralyzed muscles has long been a popular intervention for patients with Bell palsy.

Kabat rehabilitation is a type of motor control rehabilitation technique based on proprioceptive neuromuscular facilitation. Kabat technique with electrical stimulation of facial muscle is suggested to be effective in improving facial function and reducing facial disability after Bell's palsy

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis acute unilateral Bell's palsy.

Exclusion Criteria:

1. Any concurrent acute ischemia either cardiovascular or cerebrovascular disease.
2. Diabetic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
facial nerve ultrasonography | at baseline
  Thickness of facial nerve measured at the thickest part (measured by millimeters)

REFERENCES:
- [Background] Monini S, Iacolucci CM, Di Traglia M, Lazzarino AI, Barbara M. Role of Kabat rehabilitation in facial nerve palsy: a randomised study on severe cases of Bell's palsy. Acta Otorhinolaryngol Ital. 2016 Aug;36(4):282-288. doi: 10.14639/0392-100X-783. PMID 27734980